CLINICAL TRIAL: NCT05894226
Title: Functional and Sexual Outcomes After Laparoscopic Ventral Mesh Rectopexy for Complex Rectocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, consultant and lecturer of general surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2233
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Rectocele; Obstructive Defecation Syndrome
Keywords: Anterior rectocele; laparoscopic ventral mesh rectopexy
MeSH Terms: conditions — Rectocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic ventral mesh rectopexy arm (Experimental): those who were underwent laparoscopic ventral mesh rectopexy for rectocele.
  Interventions: Procedure: laparoscopic ventral mesh rectopexy

INTERVENTIONS:
Procedure: laparoscopic ventral mesh rectopexy — patients are treated by laparoscopic ventral mesh rectopexy for anterior rectocele

SUMMARY:
The ideal surgical strategy for treating complex rectocele remains a topic for debate, with the transanal, transperineal, and transvaginal approach and the abdominal approach being at conflict with one another. While the transvaginal repair is more popular among gynecologists, the trans abdominal approach has become increasingly common among colorectal surgeons, in part due to the rising demand for minimally invasive surgery.

DETAILED DESCRIPTION:
For the treatment of rectoceles and ODS in general, the laparoscopic method has recently come to light as a promising alternative.

Laparoscopic ventral mesh rectopexy (LVMR) was originally described for the management of rectal prolapse. However, It was also recommended with encouraging results for the treatment of large symptomatic rectocele.

The present study aims to evaluate the safety and efficacy of LVMR for complex rectocele.

ELIGIBILITY:
Inclusion Criteria:

* multiparous female patients.
* aged between 30 and 60 years
* who were diagnosed with complex anterior rectocele- more than 3cm after failed medical treatment- with history of either vaginal delivery or caesarian section.
* complex rectocele was one having any of the following features: size > 3 cm in diameter, associated enterocoele or internal rectal prolapse

Exclusion Criteria:

* paradoxical contraction of puborectalis muscle (anismus),
* complete external rectal prolapse
* fecal incontinence
* other benign anal conditions
* those who are unfit for surgery due to associated severe co-morbidities

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only female patients with anterior rectocele
Enrollment: 15 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
changes in the Wexner constipation score | 6 months
  improvement in constipation, if the score is decreasing this means improving

SECONDARY OUTCOMES:
sexual function changes | 6 months
  changes in the sexual function score post operative (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire score(PISQ-12). The lower the score the better the function.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided